CLINICAL TRIAL: NCT03085498
Title: Sportcheck Follow-Up: Physical Fitness, Cardiovascular and Psychosocial Health in Primary School Childen
Brief Title: Sportcheck Follow-Up
Status: Completed | Type: Observational
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Henner Hanssen, Prof. Dr. med. Henner Hanssen, University of Basel
Other Study IDs: EKNZ_258/12
Record Dates: First submitted 2017-02-28; First posted 2017-03-21 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Diseases; Childhood Obesity; Hypertension
Keywords: retinal vessels; physical activity; children; psychosocial health
MeSH Terms: conditions — Cardiovascular Diseases; Pediatric Obesity; Hypertension; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
The study resembles a four-year follow-up on the influence of physical activity and fitness, blood pressure, BMI and stress on vascular health in primary schoolchildren. It examines the predictive value of retinal vessel diameters for the development of childhood hypertension.

DETAILED DESCRIPTION:
The study aims to examine the usefulness of retinal vessel analysis in childhood cardiovascular prevention. It investigates the long-term influence of physical activity and fitness on retinal vessel diameters, blood pressure, BMI and psychosocial stress in children. The study aims to set new standards for an integrative primary prevention concept to initiate healthy ageing from childhood to adulthood.

ELIGIBILITY:
Inclusion Criteria:

* All fifth-graders of public primary schools in Basel-Stadt with an informed consent signed by their parents are included.

Exclusion Criteria:

* Fifth-graders with motor-or other disabilities that do not allow participation will be excluded.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will be designed as a four-year follow-up of the 2014 Sportcheck. All first-graders of primary schools in the canton Basel-Stadt took part in measurements of height, body weight and physical fitness during physical education lesson. From the 1255 children, 540 (43%) were allowed by their parents to join additional measurements of blood pressure and retinal vessel diameters and filled in questionnaires. In the year 2018, all fifth-graders of Basel-Stadt will be invited to take part in the same measurements as in 2014. All children will again conduct physical fitness tests and measurements of height and body weight during physical education. All children with an informed consent will participate in the same medical tests that were performed four years previously.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-07-07 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Retinal vessel diameter | Through study completion, an average of 1 year
  To assess whether physical activity and fitness changes during the four-year follow-up influence retinal vessel diameters in children

SECONDARY OUTCOMES:
Blood pressure | Through study completion, an average of 1 year
  To assess whether physical activity and fitness changes during the four-year follow-up influence blood pressure in children
Body mass index (BMI) | Through study completion, an average of 1 year
  To assess whether physical activity and fitness changes during the four-year follow-up influence BMI in children
Psychosocial stress exposure as assessed by the conflict subscale of the Family Environment Scale | Through study completion, an average of 1 year
  To assess whether physical activity and fitness changes during the four-year follow-up influence psychosocial stress in children
Health behavior as assessed by the HBSC Symptom Checklist | Through study completion, an average of 1 year
  To assess whether health behavior has changed during the four-year follow-up
Health-related quality of life as assessed by the KINDL-R questionnaire | Through study completion, an average of 1 year
  To assess whether physical activity and fitness changes during the four-year follow-up influence health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Henner Hanssen, Prof. Dr., Principal Investigator — University of Basel; Lukas Zahner, Prof. Dr., Principal Investigator — University of Basel
Locations (1):
- Bereich Sport- und Bewegungsmedizin, Abteilung Präventive Sportmedizin & Systemphysiologie, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lona G, Hauser C, Bade S, Kochli S, Infanger D, Endes K, Faude O, Hanssen H. Association of Parental Socioeconomic Status and Physical Activity with Development of Arterial Stiffness in Prepubertal Children. Int J Environ Res Public Health. 2021 Aug 3;18(15):8227. doi: 10.3390/ijerph18158227. PMID 34360513
- [Derived] Lona G, Hauser C, Kochli S, Infanger D, Endes K, Faude O, Hanssen H. Blood Pressure Increase and Microvascular Dysfunction Accelerate Arterial Stiffening in Children: Modulation by Physical Activity. Front Physiol. 2020 Dec 17;11:613003. doi: 10.3389/fphys.2020.613003. eCollection 2020. PMID 33391029